CLINICAL TRIAL: NCT02241980
Title: Survey of Patient and Physician Knowledge and Perception Regarding Medicare Part D Plan Selection
Status: Withdrawn | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stuart Beatty, Associate Professor - Clinical, Ohio State University
Other Study IDs: 2014H0191
Record Dates: First submitted 2014-09-09; First posted 2014-09-16 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Medicare Part D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medicare Part D patients: Survey
  Interventions: Other: Patient survey
- Physician Providers: Survey
  Interventions: Other: Physician survey

INTERVENTIONS:
Other: Patient survey
  Groups: Medicare Part D patients
Other: Physician survey
  Groups: Physician Providers

SUMMARY:
Evaluation of patients' methodology and ability to select an economical and ideal Medicare Part D prescription drug plan (PDP).

DETAILED DESCRIPTION:
The purpose of this project is to evaluate patients' methodology and ability to select an economical and ideal Medicare Part D prescription drug plan (PDP).

The primary objective of this project is to determine the percentage of patients who are enrolled in Medicare Part D who are currently enrolled in their ideal plan based on estimated costs.Secondary objectives are to determine:

1. The percentage of patients who have switched or considered switching their Medicare Part D PDP at any point during their enrollment
2. The most commonly used resources used by beneficiaries to aid in selection of a Medicare Part D PDP
3. The percentage of patients who reach the Medicare Part D donut hole as a result of their current plan
4. Physician perception of appropriate selection of Medicare Part D PDP among their patient panel
5. Physician perception of administrative time spent resolving medication issues related to Medicare Part D PDPs

ELIGIBILITY:
Patient Population

Inclusion Criteria:

* Patient of Martha Morehouse General Internal Medicine Clinic at the Ohio State University Wexner Medical Center
* Medicare A/B is listed as primary insurance
* Patients 65 years old or older

Exclusion Criteria:

* Patients less than the age of 65 years old
* Patients with Medicare Advantage plan

Physician Population

Inclusion Criteria:

* Physicians of Martha Morehouse General Internal Medicine Clinic at the Ohio State University Wexner Medical Center

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients of Martha Morehouse General Internal Medicine Clinic at the Ohio State University Wexner Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who are enrolled in Medicare Part D who are currently enrolled in their ideal plan based on estimated costs | Within 9 weeks of beginning survey

SECONDARY OUTCOMES:
The percentage of patients who have switched or considered switching their Medicare Part D PDP at any point during their enrollment | Within 9 weeks of beginning survey
The most commonly used resources used by beneficiaries to aid in selection of a Medicare Part D PDP | Within 9 weeks of beginning survey
The percentage of patients who reach the Medicare Part D donut hole as a result of their current plan | Within 9 weeks of beginning survey
Physician perception of appropriate selection of Medicare Part D PDP among their patient panel | Within 9 weeks of beginning survey
Physician perception of administrative time spent resolving medication issues related to Medicare Part D PDPs | Within 9 weeks of beginning survey

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Beatty, PharmD, Principal Investigator — Ohio State University
Locations (1):
- Martha Morehouse Internal Medicine Clinic at Ohio State University Wexner Medical Center, Columbus, Ohio, United States